CLINICAL TRIAL: NCT07324642
Title: A Randomized, Single-center, Single-blind, Placebo-controlled, Dose Escalation Phase 1 Clinical Trial to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Characteristics of Multiple Intravenous Infusions of KINE-101 in Healthy Adult Volunteers
Brief Title: A Phase 1 MAD Study of KINE-101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kine Sciences Co., Ltd. (Industry)
Collaborators: Chungbuk National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIDP101-CR1-002P
Record Dates: First submitted 2025-12-09; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KINE-101 (Experimental)
  Interventions: Drug: KINE-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KINE-101 — KINE-101 injection, 12.5 mg/mL, intravenous infusion once daily for 7 days under fasting conditions.
  Arms: KINE-101
Drug: Placebo — 0.9% sodium chloride, intravenous infusion once daily for 7 days under fasting conditions.
  Arms: Placebo

SUMMARY:
This is a randomized, single-center, single-blind, placebo-controlled, dose-escalation Phase 1 clinical trial designed to evaluate the safety, tolerability, pharmacokinetic, and pharmacodynamic characteristics of multiple intravenous (IV) infusions of KINE-101 in healthy adult volunteers.

The study includes three sequential cohorts with a total of 24 subjects (8 subjects per cohort; 6 assigned to KINE-101 and 2 to placebo). Subjects in the treatment groups receive KINE-101 once daily for 7 consecutive days at doses corresponding to their assigned cohort (Cohort 1: 120 mg, Cohort 2: 240 mg, Cohort 3: 360 mg). Subjects in the placebo group receive 0.9% saline under identical conditions. All subjects are admitted on Day -1, receive daily dosing from Day 1 through Day 7, and are discharged on Day 9 after completion of safety monitoring. Follow-up visits are conducted on Days 14, 21, 28, and 35. Dose escalation proceeds sequentially from the lowest-dose cohort (Cohort 1) to the highest-dose cohort (Cohort 3). Safety and tolerability data collected through Day 35 in each preceding cohort are reviewed before initiating dosing in the next higher-dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults aged 19 to 55 years
* Body weight ≥ 50.0 kg and Body Mass Index (BMI) between 18.5 and 30.0 kg/m²
* Clinically healthy with no congenital or chronic diseases requiring treatment
* Normal findings in physical examination, vital signs, 12-lead ECG, and clinical laboratory tests at screening
* Provided written informed consent and willing to comply with all study restrictions and procedures

Exclusion Criteria:

* History or presence of clinically significant hepatic, renal, cardiovascular, respiratory, neurological, hematologic, endocrine, psychiatric, or malignant diseases
* Abnormal ECG findings (QTc > 450 ms for males or > 470 ms for females; PR > 200 ms; QRS > 120 ms)
* Abnormal liver or renal function (AST, ALT, ALP, γ-GT, or total bilirubin > 2× ULN; eGFR < 60 mL/min/1.73 m²)
* Positive drug abuse test or history of substance abuse
* Abnormal vital signs at screening (SBP ≤ 90 or ≥ 150 mmHg; DBP ≤ 60 or ≥ 100 mmHg; pulse ≤ 40 or ≥ 100 bpm)
* Vaccination with live or attenuated vaccines or systemic corticosteroid use within 3 months before dosing
* Use of enzyme-inducing/inhibiting drugs, herbal medicines, or other investigational products within 1-3 months before dosing
* Donation or transfusion of blood within 3 months before dosing
* Regular alcohol consumption > 21 units/week, or inability to abstain during the study
* Current smokers (> 10 cigarettes/day) or inability to refrain from smoking during study participation
* Intake of alcohol, grapefruit, quinine, Seville orange, or caffeine-containing products within 24-72 hours before dosing and during sampling periods
* Engagement in strenuous exercise within 48 hours before dosing
* Pregnant or breastfeeding women, or men and women not using reliable contraception
* Recent COVID-19 or influenza infection or vaccination within 2 weeks before dosing
* Difficult venous access or positive alcohol breath test
* Any other condition that, in the investigator's judgment, would make the subject unsuitable for participation in the study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From Day 1 to Day 35 (End of Study visit)
  Number and percentage of subjects experiencing any treatment-emergent adverse event (TEAE) following multiple intravenous administrations of KINE-101 or placebo. Safety assessments will also include concomitant medications, physical examinations, local injection site reactions, and vital signs.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | From Day 1 (pre-dose) through Day 7 post-dose
  Maximum plasma concentration (Cmax) of KINE-101 following single and multiple doses.
Area under the plasma concentration-time curve (AUC) | From Day 1 (pre-dose) through Day 7 post-dose
  Area under the plasma concentration-time curve (AUC) of KINE-101 following single and multiple doses.
Terminal half life (t½) | From Day 1 (pre-dose) through Day 7 post-dose
  Terminal half life (t½) of KINE-101 following single and multiple doses.

OTHER OUTCOMES:
Change from baseline in serum biomarkers following KINE-101 administration | From Day 1 to Day 35 (End of Study visit)
  The change from baseline in serum biomarkers following intravenous administration of KINE-101 including IgG, IgM, IL-2, IL-6, IL-10, IL-17, IFN-gamma, MCP-1, and TGF-beta.
Change from baseline in immunophenotyping markers following KINE-101 administration | From Day 1 to Day 35 (End of Study visit)
  The change from baseline in immunophenotyping markers following intravenous administration of KINE-101 including CD4, CD25, FoxP3, CD39, CD69, LAG-3, CTLA-4, TNFR2, TIGIT, CCR5, and CXCR3.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Park, Study Director — Kine Sciences Co., Ltd.
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea

IPD SHARING:
Plan to Share IPD: No